CLINICAL TRIAL: NCT03676218
Title: Assessing Patient-reported Outcomes (PROs) and Patient-related Outcomes in Randomized Cancer Clinical Trials for Older Adults: the DATECAN-ELDERLY Initiative
Brief Title: Assessing Patient-reported & Patient-related Outcomes in Randomized Cancer Trials for Older Adults
Acronym: DATECANelderly
Status: Completed | Type: Observational
Sponsor: Institut Bergonié (Other)
Collaborators: European Organisation for Research and Treatment of Cancer - EORTC (Network); International Society of Geriatric Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: IB2016-DATECAN-elderly
Record Dates: First submitted 2018-09-17; First posted 2018-09-18 (Actual); Results first posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Cancer
Keywords: Cancer; Elderly; Randomized controlled trial; Endpoint; Consensus
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elderly cancer patients: Experts involved in the experts' panel for providing recommandations for the definitions of time to event outcomes to be used in randomized trials for older patients with cancer
  Interventions: Other: Elderly cancer patients

INTERVENTIONS:
Other: Elderly cancer patients — No intervention: Panel of international experts to provide definition of survival endpoints to be used in randomized controlled trials to assess treatment efficacy.

SUMMARY:
As older adults with cancer are underrepresented in randomized clinical trials (RCT), there is limited evidence on which to rely for treatment decisions for this population. Commonly used RCT endpoints for the assessment of treatment efficacy are more often tumor-centered (e.g., progression-free survival). These endpoints may not be as relevant for the older patients who present more often with comorbidities, non-cancer-related deaths, and treatment toxicity. Moreover, their expectation and preferences are likely to differ from younger adults.

The DATECAN-ELDERLY initiative combines a broad expertise, in geriatric oncology and clinical research, with interest in cancer RCT that include older patients with cancer. In order to guide researchers and clinicians coordinating cancer RCT involving older patients with cancer, the experts reviewed the literature on relevant domains to assess using patient-reported outcomes (PRO) and patient-related outcomes, as well as available tools related to these domains.

Domains considered relevant by the panel of experts when assessing treatment efficacy in RCT for older patients with cancer included functional autonomy, cognition, depression and nutrition. These were based on published guidelines from international societies and from regulatory authorities as well as minimum datasets recommended to collect in RCT including older adults with cancer. In addition, health-related quality of life, patients' symptoms, and satisfaction were also considered by the panel. With regards to tools for the assessment of these domains, we highlighted that each tool has its own strengths and limitations, and very few had been validated in older adults with cancer. Further studies are thus needed to validate these tools in this specific population and define the minimum clinically important difference to use when developing RCTs in this

DETAILED DESCRIPTION:
In cancer randomized controlled trials (RCT), the validated and most objectively defined evaluation criterion is overall survival (OS - delay between randomization and death). Therapeutic progress, the current context of strategic trials, and the multiplication of lines of treatment have resulted in the necessity to identify evaluation criteria other than OS, which can be observed more frequently and sooner. Endpoints such as progression-free survival (PFS) or disease-free survival (DFS) are commonly used instead of OS in RCT. The priority for patients, however, is to live longer or better, and ideally both, which raises the question as to the suitability of these tumor-specific endpoints to assess the benefit/risk balance associated to a new therapy in elderly patients with cancer. Older patients may die from causes other than cancer, and relapse does not necessarily shorten survival. Instead, cancer therapy can sometimes cause severe acute or chronic toxicities and affect functional status or health-related quality of life (HRQoL), and as such these patient-centered outcomes (e.g. autonomy, quality of life) should be given more attention. On the basis of these considerations, OS may not be the most appropriate outcome to measure treatment benefit in the elderly cancer population.

Geriatric oncology experts and task forces including the International Society of Geriatric Oncology, the European Organization for Research and Treatment Cancer (EORTC) and the DIALOG research group (Dialogue Intergroupe pour la personnALisation de la prise en charge en OncoGériatrie), have acknowledged the heterogeneity of primary endpoints used in RCT conducted in elderly cancer patients. This heterogeneity, in terms of dimension (tumor-centered outcomes, patient-centered outcomes including autonomy, nutrition, etc.) and definitions limits the comparison of results across trials. In addition, this can make the design of trials particularly complex since estimation of sample size is usually based on results from past trials. Acknowledging the specificities of the elderly population, the DATECAN-Elderly project is aimed at providing guidelines for the definition of efficacy endpoints that will permit to assess new treatments/interventions in this population.

The DATECAN-Elderly project is a continuation of the development of guidelines within the DATECAN initiative (Definition for the Assessment of Time-to-event Endpoints in CANcer trials). This international initiative was launched in 2009 to elaborate standardized definitions for survival endpoints in RCT, based on a rigorous and validated consensus methodology. This work has resulted in the publication of guidelines to define time-to-event endpoints to be used in randomized trials for specific cancer sites: sarcomas, pancreas, breast, and other. These guidelines however were not developed for the elderly cancer patients. Events specifically accounted for included exclusively tumor-oriented events (e.g. local, regional, metastatic progressions, or deaths due to various causes).

DATECAN-Elderly guidelines will be developed in cooperation with many experts in the field of geriatric oncology and clinical trials from different scientific backgrounds (medical oncologists, geriatricians, biostatisticians, etc.) and groups/societies (DIALOG, SIOG, EORTC, etc.), favouring the acceptability of the resulting recommendations. R

Results of the DATECAN-Elderly project are expected to address the heterogeneity regarding efficacy endpoints used as primary endpoints in elderly cancer trials. Providing definitions for endpoints should lead to the evaluation of treatment more consistent with patient's experiences and expectations about treatment outcome. Overall, the project should help provide trials' results which are more relevant for the elderly patients, improves the recruitment of elderly patient in RCT, and finally enhance trials' comparison and design.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients with cancer

Exclusion Criteria:

* Individual patient data unavailable

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: No patient will be included.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carine Bellera, PhD, Principal Investigator — Institut Bergonié
Locations (1):
- Institut Bergonié, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Galvin A, Soubeyran P, Brain E, Cheung KL, Hamaker ME, Kanesvaran R, Mauer M, Mohile S, Montroni I, Puts M, Rostoft S, Wildiers H, Mathoulin-Pelissier S, Bellera C. Assessing patient-reported outcomes (PROs) and patient-related outcomes in randomized cancer clinical trials for older adults: Results of DATECAN-ELDERLY initiative. J Geriatr Oncol. 2024 Jan;15(1):101611. doi: 10.1016/j.jgo.2023.101611. Epub 2023 Sep 9. PMID 37679204

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants Involved in the Panel of International Experts: Experts involved in the panel of experts for providing recommandations for the definitions of time to event outcomes to be used in randomized trials for older patients with cancer
  No intervention: Panel of international experts to provide definition of survival endpoints to be used in randomized controlled trials to assess treatment efficacy.
Period: Overall Study
Arm/Group | Participants Involved in the Panel of International Experts
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 14 experts participated in the panel
Arm/Group | Participants Involved in the Panel of International Experts
Number analyzed (Participants) | 14
Age, Customized [Count of Participants; unit: Participants]
  older than 18 years | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 5
  United Kingdom | 1
  Netherlands | 1
  Singapore | 1
  Belgium | 2
  United States | 1
  Italy | 1
  Norway | 1
  Canada | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Domains Considered Relevant by the Panel of Experts When Assessing Treatment Efficacy in Randomized Cancer Trials for Older Patients With Cancer
Description: The domains were selected by the panel of experts based on the published guidelines (scientific societies, regulatory authorities, minimum datasets).
  Domains included functional autonomy, cognition, depression and nutrition. In addition, health-related quality of life, patients' symptoms, and satisfaction were also considered by the panel.
Time Frame: 1 year after the consitution of the panel of experts
Measure: Number; unit: geriatric domains
Arm/Group | Participants Involved in the Panel of International Experts
Number analyzed (Participants) | 14
geriatric domains | 7

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Participants Involved in the Panel of International Experts
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2015-07-18): https://cdn.clinicaltrials.gov/large-docs/18/NCT03676218/Prot_000.pdf